CLINICAL TRIAL: NCT07375095
Title: Effect of BH-SLP-001 Sleep Supplement on Sleep Parameters in Menopausal Women: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: A Study of a Sleep Supplement to Improve Sleep in Women Going Through Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bonafide Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00073864
Record Dates: First submitted 2025-11-24; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Sleep Disturbance
Keywords: Menopause; Perimenopause; Postmenopause; Sleep Disturbance; Sleep Quality; Sleep Onset Latency; Wake After Sleep Onset; Nighttime Awakenings; Women's Health
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: A two-arm, randomized, double-blind, placebo-controlled parallel assignment in which participants were allocated to either the dietary supplement or placebo group and remained in the same group for the duration of the 21-day intervention. All study procedures were conducted virtually.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study used a double-blind design in which participants, investigators, care providers, and outcomes assessors were unaware of group assignment. The supplement and placebo were matched in appearance, packaging, and administration instructions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Supplement Arm (Experimental): Participants received the dietary sleep supplement once daily for 21 days. The product was taken 60 minutes before bedtime during the intervention period. All dosing and study activities were conducted virtually.
  Interventions: Dietary Supplement: Sleep Supplement
- Placebo Arm (Placebo Comparator): Participants received a placebo matched in appearance and dosing schedule to the supplement. The placebo was taken once daily, 60 minutes before bedtime, for 21 days. All dosing and study activities were conducted virtually.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Sleep Supplement — A daily dietary sleep supplement taken once per day for 21 days.
  Arms: Dietary Supplement Arm
Drug: Placebo — A placebo matched in appearance and dosing schedule to the sleep supplement, taken once per day for 21 days.
  Arms: Placebo Arm

SUMMARY:
This study evaluated whether a daily dietary sleep supplement could improve sleep in women aged 40 to 65 who experience moderate sleep disturbances during menopause. Participants were randomly assigned to take either the supplement or a placebo for about three weeks. All study visits were conducted virtually. Sleep was assessed through daily diaries and weekly questionnaires measuring sleep quality, nighttime awakenings, daytime alertness, and mood. The study's goal was to compare changes between the supplement and placebo groups and to assess safety and tolerability during the study period.

DETAILED DESCRIPTION:
This study was a randomized, double-blind, placebo-controlled, parallel-group clinical trial conducted to evaluate the effects of a dietary sleep supplement on subjective sleep disturbance, sleep-related impairment, and related sleep parameters in perimenopausal and postmenopausal women with moderate sleep complaints.

Participants were enrolled remotely and randomized in a 1:1 ratio to receive either the investigational dietary supplement or a matching placebo. Randomization was performed using a blinded allocation scheme, and blinding was maintained for participants and all study personnel involved in participant management, data collection, and outcome assessment. Study products were physically and visuallyishable to preserve masking throughout the study.

Following electronic informed consent, participants completed a screening phase conducted via virtual visit, during which baseline sleep disturbance and medical history were assessed to confirm eligibility. Eligible participants then entered a run-in period of approximately seven days, during which they completed daily electronic sleep diaries to establish baseline sleep patterns and to familiarize themselves with study procedures. No study product was consumed during the run-in period.

After completion of the run-in phase, participants initiated the intervention period (Day 1) and self-administered the assigned study product once daily for 21 ± 3 days. The investigational product was administered orally approximately 60 minutes before bedtime, and participants randomized to placebo followed an identical dosing schedule.

Throughout the intervention period, participants completed daily electronic sleep diaries and periodic electronic questionnaires assessing changes in sleep disturbance, sleep-related impairment, overall sleep quality, and daytime functioning. Assessments were collected at baseline and at regular intervals during the dosing period, consistent with the protocol-defined schedule of activities. At the end-of-study visit, participants completed a product experience questionnaire evaluating usability and overall experience with the study product.

All study visits and assessments were conducted remotely. Safety and tolerability were monitored throughout the study through participant self-report and scheduled virtual check-ins. Adverse events were collected, assessed for severity and relatedness, and followed through resolution in accordance with protocol-defined safety monitoring procedures.

Each participant's total duration of participation was approximately four to five weeks, including screening, run-in, intervention, and end-of-study assessments. The study was designed to characterize the short-term effects, safety, and tolerability of a dietary sleep supplement in menopausal women experiencing moderate sleep disturbance under fully remote study conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women who are 40 to 65 years of age (inclusive).
2. Have a body mass index (BMI) between 18.5 to 34.9 kg/m2 (inclusive).
3. PROMIS SD SF T-Score Cut Point ≥ 60 (equivalent to a raw score of 30).
4. Women enrolled in this research study may be of perimenopausal, (12 or more months without a menstrual period) or post-menopausal status.

   1. Post-menopause defined as the last natural menstrual period (LNMP) completed at least 12 months prior to screening.
   2. Perimenopause defined as women who complained of irregular menstrual cycle in the past 12 months, with a forward or postponed cycle more than 7 days.

   i. At least 2 cycles were missing during the past 12 months or reported menopause for at least 60 days.
5. In good general health (no active or uncontrolled diseases or conditions) and able to consume the study product.
6. Agree to refrain from treatments listed in Section 12.4 in the defined timeframe.
7. Has stable access to Wi-Fi and an iPhone or Android device.
8. Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion Criteria:

1. Individuals who are lactating, pregnant, or planning to become pregnant during the study.
2. Perimenopausal women who are sexually active will be required to specify contraceptive method or be excluded.
3. Currently incarcerated prisoners.
4. Currently enrolled in a different clinical trial.
5. Previous use of SAM-e, PG, GABA, Theanine, and/or Magnesium (unless in a multivitamin) within 3 months prior to screening.
6. Use of any treatment for sleep symptoms or other concomitant treatments listed in Section 12.4.
7. Taking blood thinners within the last 2 weeks. Further details may be found in Section 12.4.
8. Have a known sensitivity, intolerability, or allergy to any of the study products or their excipients.
9. Received a vaccine for COVID-19 in the two weeks prior to screening or during the study period, current COVID-19 infections, or currently have the post-COVID-19 condition as defined by World Health Organization (WHO) (i.e., individuals with a history of probable or confirmed SARS-CoV-2 infection, usually three months from the onset of COVID-19 with symptoms that last for at least two months and cannot be explained by an alternative diagnosis).
10. Have a positive medical history of heart disease, renal disease, hepatic impairment, or active systemic infection (e.g., Lyme disease, TB, HIV).
11. History of cancer (except localized skin cancer without metastases) within two (2) years prior to screening.
12. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential subject at risk because of participation in the study or influence the results or the potential subject's ability to participate in the study.
13. History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs (i.e., Crohn's disease, short bowel, acute or chronic pancreatitis, or pancreatic insufficiency).
14. Participant has an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g., dysphagia) and digestion (e.g., known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea).
15. Major surgery in three months prior to screening or planned major surgery during the study.
16. Currently diagnosed with depression by a doctor or physician.
17. Have been or currently diagnosed with bipolar disorder by a doctor or physician.
18. History of epilepsy or taking epileptic medications.
19. Presence of sleep disorders that have been diagnosed by a doctor or physician.
20. Currently using any sleep device (e.g., nebulizer machine, sleep apnea masks, continuous positive airway pressure (CPAP)) to improve sleep.
21. Recent shift work, night work, or frequent travel to different time zones in the past month, which, in the opinion of the investigator, may adversely affect the participant's sleep quality.
22. Consumption of more than 400 mg of caffeine per day.
23. History of alcohol or substance abuse in the last 5 years.
24. Report ≥ 5 night sweats per week.
25. Report ≥20 hot flashes per week.
26. Have animals that frequently cause sleep disturbances
27. Have partners who regularly disturb their sleep
28. Have young children or infants who frequently require caregiving responsibilities and disturb sleep
29. Planned travel during the study period that, in the opinion of the investigator, may negatively influence the participant's sleep.
30. Any other active or unstable medical conditions or use of medications/supplements/ therapies that, in the opinion of the investigator, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant. Note: screened participants with infections would be eligible to participate four weeks after completing their treatment (wash-out period).

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-04-07 (Actual); Study Completion 2024-04-07 (Actual)

PRIMARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System (PROMIS®) Sleep Disturbance Short Form 8b T-score | Day -7 (run-in baseline) to Day 21 (±3 days)
  Change from baseline in the Patient-Reported Outcomes Measurement Information System (PROMIS®) Sleep Disturbance Short Form 8b T-score, a validated patient-reported outcome measure assessing perceived sleep quality, difficulty falling or staying asleep, and overall sleep satisfaction over the prior 7 days. The PROMIS Sleep Disturbance Short Form 8b yields raw scores ranging from 8 to 40, which are converted to standardized T-scores ranging from 28.9 to 76.5. Higher T-scores indicate greater sleep disturbance (worse sleep outcomes).
Responder Rate for Patient-Reported Outcomes Measurement Information System (PROMIS®) Sleep Disturbance Short Form 8b | Day -7 (run-in baseline) to Day 21 (±3 days)
  Responder rate defined as the proportion of participants achieving a clinically meaningful improvement in sleep disturbance, as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS®) Sleep Disturbance Short Form 8b T-score. The PROMIS Sleep Disturbance Short Form 8b yields raw scores ranging from 8 to 40, corresponding to standardized T-scores ranging from 28.9 to 76.5, with higher scores indicating greater sleep disturbance (worse sleep outcomes). Responders were defined as participants who experienced a decrease of ≥8 points in the PROMIS Sleep Disturbance T-score from baseline, consistent with the established minimal clinically important difference (MCID) for this measure.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS®) Sleep-Related Impairment Short Form 8a T-score | Day -7 (run-in baseline) to Day 21 (±3 days)
  Change from baseline in the Patient-Reported Outcomes Measurement Information System (PROMIS®) Sleep-Related Impairment Short Form 8a T-score, a validated patient-reported outcome measure assessing daytime alertness, sleepiness, fatigue, and functional impairment related to sleep over the prior 7 days. The PROMIS Sleep-Related Impairment Short Form 8a yields raw scores ranging from 8 to 40, which are converted to standardized T-scores ranging from 30.0 to 80.1. Higher T-scores indicate greater sleep-related impairment (worse daytime functioning).
Responder Rate for Patient-Reported Outcomes Measurement Information System (PROMIS®) Sleep-Related Impairment Short Form 8a | Day -7 (run-in baseline) to Day 21 (±3 days)
  Responder rate defined as the proportion of participants achieving a clinically meaningful improvement in sleep-related impairment, as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS®) Sleep-Related Impairment Short Form 8a T-score. The PROMIS Sleep-Related Impairment Short Form 8a yields raw scores ranging from 8 to 40, corresponding to standardized T-scores ranging from 30.0 to 80.1, with higher scores indicating greater sleep-related impairment (worse daytime functioning). Responders were defined as participants who experienced a decrease of ≥6.5 points in the PROMIS Sleep-Related Impairment T-score from baseline, based on the 95% reliable change index (RCI), representing a magnitude of change exceeding measurement error and consistent with clinically meaningful improvement in similarly aged adults with sleep-related impairment.

SECONDARY OUTCOMES:
Change in Sleep Quality as Measured by a Visual Analog Scale (VAS) | Day -7 (run-in baseline) to Day 21 (±3 days)
  Change from baseline in self-reported sleep quality measured using a visual analog scale (VAS) ranging from 0 to 100, where lower scores indicate better sleep quality and higher scores indicate poorer sleep quality or satisfaction. Improvement in sleep quality is reflected by a decrease in VAS score from baseline.
Change in Total Sleep Time (TST) | Day -7 (run-in baseline) to Day 21 (±3 days)
  Change from baseline in total nightly sleep duration, measured in minutes, as recorded in daily morning sleep diaries. Higher values indicate longer total sleep time, with increases from baseline reflecting improvement in sleep duration.
Change in Sleep Efficiency | Day -7 (run-in baseline) to Day 21 (±3 days)
  Change in sleep efficiency calculated from daily diary entries as the ratio of total sleep time to time in bed.
Change in Sleep-Onset Latency (SOL) | Day -7 to Day 21 (±3 days)
  Change from baseline in sleep-onset latency, measured in minutes, defined as the time required to fall asleep after attempting to sleep, as recorded in daily morning sleep diaries. Lower values indicate shorter sleep-onset latency, with decreases from baseline reflecting improvement in sleep initiation.
Change in Difficulty Falling Asleep as Measured by a Visual Analog Scale (VAS) | Day -7 (run-in baseline) to Day 21 (±3 days)
  Change from baseline in self-reported difficulty falling asleep measured using a visual analog scale (VAS) ranging from 0 to 100, where lower scores indicate less difficulty falling asleep and higher scores indicate greater difficulty. Improvement is reflected by a decrease in VAS score from baseline.
Change in Wake After Sleep Onset (WASO) | Day -7 to Day 21 (±3 days)
  Change from baseline in wake after sleep onset (WASO), measured in minutes, defined as the total time spent awake after initially falling asleep, as recorded in daily morning sleep diaries. Lower values indicate less wake time after sleep onset, with decreases from baseline reflecting improvement in sleep maintenance.
Change in Number of Spontaneous Nighttime Awakenings | Day -7 (run-in baseline) to Day 21 (±3 days)
  Change from baseline in the number of spontaneous nighttime awakenings, measured as a count per night, as recorded in daily morning sleep diaries. Lower values indicate fewer awakenings, with decreases from baseline reflecting improvement in sleep continuity.
Change in Sleep Disturbance as Measured by a Visual Analog Scale (VAS) | Day -7 (run-in baseline) to Day 21 (±3 days)
  Change from baseline in self-reported sleep disturbance measured using a visual analog scale (VAS) ranging from 0 to 100, where lower scores indicate less perceived sleep disturbance and higher scores indicate greater disturbance. Improvement is reflected by a decrease in VAS score from baseline.
Change in Number of Nocturia Episodes | Day -7 (run-in baseline) to Day 21 (±3 days)
  Change from baseline in the number of nocturia episodes per night, measured as a count, defined as the number of times a participant awakened to use the restroom during the night, as recorded in daily morning sleep diaries. Lower values indicate fewer nocturnal bathroom visits, with decreases from baseline reflecting improvement in sleep maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Trisha VanDusseldorp, PhD, Principal Investigator — Bonafide Health, LLC
Locations (1):
- Bonafide Health, LLC, Harrison, New York, United States

IPD SHARING:
Plan to Share IPD: No